CLINICAL TRIAL: NCT04726865
Title: Effects of COVID-19 Pandemic on Medical Students in Jordanian Universities: A Multi-center Cross-sectional Study
Brief Title: COVID-19 Pandemic and Medical Students
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Collaborators: Aysha Alkhayat (Unknown); Mariam Aljweesri (Unknown); Reem Alharbi (Unknown); Zahraa Aljazzaf (Unknown)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, Jordan University Hospital
Other Study IDs: Jordan Universities
Record Dates: First submitted 2021-01-25; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: the Effect of COVID-19 Pandemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Naser Al-Husban — voluntary completion of an online questionnaire

SUMMARY:
Little is known about changes in levels of academic, financial, psychological, & hygienic impact on medical students during this pandemic.

DETAILED DESCRIPTION:
this is a cross-sectional, questionnaire-based study. It is conducted on a random targeted sample of medical students at medical schools in Universities of Jordan, classified by their academic years (from the 1st to the 6th academic year). A score of 10 points was constructed to reflect the perspective about the items in each group of variables. SPSS version 25.0 was used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Medical students in the basic and clinical years

Exclusion Criteria:

* Inability to complete the questionnaire

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Medical students
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
psychological stress and academic results | 2 months
  e- questionnaire will be completed by students. The questionnaire was built through google forms (without relying on pre-existing ones) and was made available in Arabic.

CONTACTS AND LOCATIONS:
Overall Officials: Naser U Al-Husban, Principal Investigator — The University of Jordan
Locations (1):
- Al-Husban University Naser, Amman, Jordan